CLINICAL TRIAL: NCT05129254
Title: A Pilot Study Evaluating the Safety and Efficacy of a Fractionated Thulium Laser and Topical Platelet Rich Plasma vs. Platelet Rich Plasma Injection for the Treatment of Male Androgenetic Alopecia
Brief Title: Thulium Laser and Topical Platelet Rich Plasma (PRP) vs. PRP Injection for the Treatment of Male Androgenetic Alopecia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not initiated.
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-13642
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Androgenetic Alopecia
Keywords: alopecia; laser; platelet rich plasma; male pattern hair loss
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Intervention Model Description: To compare the efficacy of laser to improve delivery of topical platelet rich plasma (PRP) to promote hair growth, the investigators will employ a randomized, unblinded, baseline-controlled study design. There will be two parallel treatment arms in the study. The first arm will enroll six participants to receive thulium laser and topical PRP. The second arm will enroll six participants to receive PRP injection alone. Total participants enrolled will be twelve (12). There will be a total of 8 study visits (4 treatment and 4 follow-up) lasting 16 months.
  Each participant will receive an initial series of 4 treatments, either laser + topical PRP or PRP injection alone once a month for the first 4 months (month 1, 2, 3, 4). Thereafter, patients will be followed at 3-month intervals at month 7, 10, 13, and 16.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thulium laser (1927nm) and post-treatment topically administered platelet rich plasma (PRP) (Experimental): All participating subjects will serve as their own baseline control and will receive treatment of their androgenetic alopecia with LaseMD, a 1927nm Fractionated Thulium laser and post-treatment topically applied autologous platelet rich plasma at monthly intervals for a total of 4 treatment. The total duration of laser application, venipuncture, PRP preparation, and topical administration will take approximately 30 minutes. Post-treatment surveillance: The subject will be observed in the clinic under direct supervision of the treating physician for any post-treatment side-effects for up to 15 minutes.
  Interventions: Device: Fractionated Thulium laser; Procedure: Autologous Platelet Rich Plasma Topical Application
- Platelet rich plasma injection (Experimental): All participating subjects will serve as their own baseline control and will receive treatment of their androgenetic alopecia with autologous platelet rich plasma injection at monthly intervals for a total of 4 treatment. The total duration of venipuncture, PRP preparation, and injection will take approximately 15 minutes. Post-treatment surveillance: The subject will be observed in the clinic under direct supervision of the treating physician for any post-treatment side-effects for up to 15 minutes.
  Interventions: Procedure: Autologous Platelet Rich Plasma Injection

INTERVENTIONS:
Device: Fractionated Thulium laser — For this study, the investigators will use non-ablative fractional Thulium laser (1927 nm), provided by LaseMD, (Lutronic, Inc, USA). The non-ablative fractionated treatments with minimal downtime provide synergistic benefit of minimizing tissue damage while improving treatment tolerance and efficiency. The laser works by creating micro-channels in the dermis of the pilosebaceous unit, while leaving bridges of untouched tissue for improved permeability, faster healing, and enhanced delivery of topical treatments. The parameters of the laser will be set according to optimal operation protocol and in accordance with guidelines set forth by LaseMD. More than one affected area of the scalp may be treated per session. Each laser treatment will take approximately 10 to 15 minutes per subject. Pretreatment preparation will consist of cleaning the affected area of the scalp with antiseptic, either 70% ethanol or 3% hydrogen peroxide.
  Other Names: LaseMD Lutronic Laser
  Arms: Thulium laser (1927nm) and post-treatment topically administered platelet rich plasma (PRP)
Procedure: Autologous Platelet Rich Plasma Injection — Platelet rich plasma (PRP) will be collected from participant in accordance with FDA section 21CFR640.34 regulation on collection and preparation of PRP. The collected blood will be processed according to manufacturer protocol to obtain PRP, which will be injected with a syringe and needle subcutaneously into the participant's scalp.
  Arms: Platelet rich plasma injection
Procedure: Autologous Platelet Rich Plasma Topical Application — Platelet rich plasma (PRP) will be collected from participant in accordance with FDA section 21CFR640.34 regulation on collection and preparation of PRP. The collected blood will be processed according to manufacturer protocol to obtain PRP, which will be applied topically with a syringe to one or more affected areas on the participant's scalp that were previously treated with thulium laser.
  Arms: Thulium laser (1927nm) and post-treatment topically administered platelet rich plasma (PRP)

SUMMARY:
The objective of this clinical study is to compare the safety and efficacy of a laser and topically applied platelet-rich plasma vs. platelet rich plasma injection in the treatment of male-pattern hair loss. Participating subjects will receive up to four (4) monthly treatments and will have a 12 month follow-up period.

DETAILED DESCRIPTION:
This is a single institution, open-label, baseline-controlled, prospective study evaluating the use of a non-ablative fractionated thulium laser and topical autologous platelet-rich plasma (PRP) vs. PRP injection for the treatment of male androgenetic alopecia (MAA). Given that this is a feasibility study, the investigators do provide formal sample size calculations. The findings of the study will inform that effect size associated with the treatment under study, which will inform the sample size (and power) calculations of a full, large-scale study. For this feasibility study, the investigators conservatively estimated the number of eligible patients that can reasonably enroll in the study time frame. Over the course of 1 year, the investigators typically see 50 patients with this condition annually. Of those, the investigators anticipate 25-50% would be eligible and agree to participate in the study. Given this, the investigators reasonably believe the enrollment will be 12 male subjects, ≥ 18 years of age at time of signed informed consent, of whom 6 will be randomized to receive laser + topical PRP and 6 to receive PRP injection. Follow-up visits are planned for months 7, 10, 13, and 16. Standardized photography, hair density measurement of the treated scalp areas will be recorded Pre and Post Treatment at each visit. Measurement outcomes will be compared to baseline. During the initial visit, subjects who meet the study's eligibility criteria will receive the first treatment after signing informed consent form.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male, ≥ 18 years of age at time of informed consent, seeking treatment for hair loss.
* Subject must voluntarily sign and date an IRB approved informed consent form
* Subjects with diagnosis of androgenetic alopecia with hair loss recorded over the past 6 months. (Norwood Hamilton Class 3-4 for males)
* Able to read, understand and voluntarily provide written informed consent.
* Subject is determined to be healthy, non-smoker who agrees not to make any changes to their daily hair treatment regime during the study.
* Subjects able and willing to comply with the treatment protocol and follow-up schedule and requirements.
* Understands and accepts the obligation not to undergo any other procedures in the areas to be treated through the follow-up period.

Exclusion Criteria:

* Subjects does not have the capacity to consent to the study
* Subject has other types of alopecia of the scalp (i.g., alopecia areata, scarring alopecia)
* Use of minoxidil or 5-alpha reductase inhibitors (i.e., finasteride, dutasteride) 3 months prior to screening date.
* Any medical condition that in the consideration of the investigator, would present an increased risk of a photosensitivity reaction to the subject.
* Any previous surgical procedure in the treatment area in the past 12 months, or major surgery in the last 6 months.
* History of immunosuppression/immune deficiency disorders (including AIDS and HIV infection), and/or any history of systemic chemotherapy for prior 12 months.
* History or current use of the following prescription medications:

  i. Immunosuppressive medications/biologics, 6 months prior to and during the study ii. Accutane or other systemic retinoids within the past twelve months
* Smoking or vaping in the past 12 months.
* History of hyperlipidemia, diabetes mellitus, hepatitis, or bleeding disorders.
* History of major depressive disorders or endocrine disorders including but not limited to; hypothyroidism, Hashimoto's thyroiditis, or hyperthyroidism.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male with biopsy proven diagnosis of androgenetic alopecia
Enrollment: 0 (Actual)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects with score of 2 or 3 on Clinician Global Aesthetic Improvement (CGAIS) scale at month 7 follow-up. | 7 months
  Clinician Global Aesthetic Improvement Scale (CGAIS) is a Likert scale, ranging from "greatly decreased (-3)" hair growth to "greatly increased (+3)" hair growth.
  Greatly decreased (-3) Moderately decreased (-2) Slightly decreased (-1) No change (0) Slightly increased (+1) Moderately increased (+2) Greatly increased (+3)
  Based on a live assessment of the subject while referring to the subject's pre-treatment scalp photographs, the clinician will make an assessment of post-treatment hair growth.
Percentage of subjects with score of 2 or 3 on Subject Global Aesthetic Improvement at month 7 follow-up. | 7 months
  Subject Global Aesthetic Improvement Scale (SGAIS) is a Likert scale, ranging from "greatly decreased (-3)" hair growth to "greatly increased (+3)" hair growth.
  Greatly decreased (-3) Moderately decreased (-2) Slightly decreased (-1) No change (0) Slightly increased (+1) Moderately increased (+2) Greatly increased (+3) Subjects will be given a hand mirror for self-assessment of post-treatment hair growth compared to subject's pre-treatment scalp photographs.

SECONDARY OUTCOMES:
Percentage of subjects with score of 2 or 3 on Patient Satisfaction Questionnaire at month 7 follow-up. | 7 months
  Patient Satisfaction Questionnaire will use Lickert scale, ranging from "greatly decreased (-3)" to "greatly increased (+3)".
  Greatly decreased (-3) Moderately decreased (-2) Slightly decreased (-1) No change (0) Slightly increased (+1) Moderately increased (+2) Greatly increased (+3)
  The seven point Lickert scale will apply to following patient satisfaction questions:
  Please choose the option that better represents the change in how your hair looks OVERALL in the area treated? Please choose the option that better represents the change in your hair THICKNESS in the area treated? Please choose the option that better represents the change in your hair SHEDDING/LOSS in the area treated? Please choose the option that better represents the change in your hair DARKNESS in the area treated.
Reported pain score on Numeric Rating Scale for Pain for first 4 months during treatment | 4 months
  The Numeric Rating Scale for Pain is an 11-point scale scored from 0-10, with 0 = no pain, 5 = moderate pain, and 10 = worst possible pain. Subjects select a value that is most in line with the intensity of their pain experienced during and after treatment with Thulium Laser and topical platelet rich plasma or platelet rich plasma injection. The NRS pain questionnaire will be given to participants to complete for each treatment for the first 4 months of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Kseniya Kobets, MD, Principal Investigator — Montefiore Medical Center